CLINICAL TRIAL: NCT01797107
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Determine the Effect of Azasite on Corneal Surface Irregularity in Subjects With Meibomian Gland Dysfunction
Brief Title: Study to Determine the Effect of Azasite on Corneal Surface Irregularity
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Philadelphia Eye Associates (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 40958
Record Dates: First submitted 2013-01-30; First posted 2013-02-22 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2015-04

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Meibomian gland dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment eye (Experimental): Azasite (azithromycin ophthalmic 1%) twice a day for 2 days followed by nightly for 4 weeks
  Interventions: Drug: Azasite
- Durasite (Placebo Comparator): Vehicle of Azasite used as placebo
  Interventions: Drug: Azasite

INTERVENTIONS:
Drug: Azasite — Patients will be given 1 drop twice a day for 2 days followed by 1 drop nightly for 4 weeks.
  Other Names: Azithromycin ophthalmic 1%

SUMMARY:
The purpose of this study is to evaluate the effect of Azasite on patients with corneal surface irregularity (meibomian gland dysfunction).

DETAILED DESCRIPTION:
This will be a single-center, randomized, vehicle-controlled, double-masked, clinical trial comparing a four week course of Azasite (azithromycin ophthalmic 1%) to vehicle (Durasite®) in patients with MGD-related evaporative dry eye. All patients will be evaluated at screening, baseline, two weeks, four weeks, and six weeks.

The primary outcome measure will be improvement, as compared to baseline, in corneal irregularity as measured by a topographically-derived value, the Corneal Irregularity Measurement (CIM). Secondary outcome measures will be a global symptom score, tear film break up time, meibomian gland secretion characteristics, best-corrected distance visual acuity, corneal staining, axial topography based astigmatism patterns, and IOL Master keratometry.

We will enroll 60 eyes of 30 patients, and each patient will be randomly assigned to receive Azasite in one eye and vehicle (Durasite®) in the fellow eye.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent prior to enrollment in study
* Patient ability to follow study instructions and comply with all study protocols
* Corneal irregularity measurement (CIM) > 1.7 in both eyes
* Non-atrophic meibomian gland dysfunction (MGD) as defined by abnormal meibomian expression in at least 2 meibomian glands of the eyelids of each eye
* At least two symptoms of at least moderate severity (≥ grade 2, 0 to 3 scale) as defined in the MGD Global Symptom Score (Itching, Foreign-body sensation, Dryness, Burning, Lid swelling)
* Tear film break up time < 10 seconds
* Schirmer with anesthesia > 5 mm
* Best corrected distance visual acuity (BCDVA) > 20/100

Exclusion Criteria:

* Cicatricial or atrophic meibomian gland dysfunction (MGD)
* Any corneal disease or scar involving the central 6 mm, including epithelial basement membrane dystrophy, Salzmann nodular degeneration, recurrent erosions, keratoconus or ectasia
* Use of azithromycin or doxycycline within 1 month of screening
* Topical ocular antibiotic, anti-histamines, allergy, or steroid medication within 2 weeks of baseline (a 2 week washout after screening will be allowed)
* Topical prostaglandin analogue use within 30 days of study
* The anticipated use of any drops, gels or ointments during the study period outside of the study protocol
* Use of eye make-up during study period
* Active ocular infection or inflammation
* History of herpetic eye disease or neurotrophic keratitis
* Lid pathology (except MGD or blepharitis) that the examiner feels may affect the ocular surface
* Significant conjunctival scars (ex. h/o SJS)
* Pterygium
* Lacrimal punctal occlusion within 2 months of screening
* Ocular surgery within 1 year of screening
* Monocular patients
* Pregnant, breast-feeding, or sexually active females not using contraception
* Uncontrolled systemic disease
* Presence of any disease (medical or ocular) that, in the opinion of the investigator, may interfere with the study's safety or interpretation
* Known allergy to the study medication or its components
* Current enrollment in an investigational drug or device study within 30 days of screening for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in Corneal Irregularity Measurement | 4 weeks
  Topographically defined corneal smoothness as compared to baseline measurement at day 0

SECONDARY OUTCOMES:
Global symptoms score | 2,4 and 6 weeks
  0-3 score of itching, foreign body sensation, dryness, burning and swelling as compared to baseline measurement at day 0
Meibomian gland secretion characteristics | 2, 4 and 6 weeks
  Meibum secretions of the eyelids will be assessed at each visit by pressing on the lower or upper lid (with a finger) until excretions are seen from at least 2 meibomian glands. The following scale, based on a scale in a study by Mathers et al (Mathers et al. Meibomian Gland Dysfunction in Chronic Blepharitis. Cornea .1991;10(4): 277-285.) will be used:
  NE= <2 glands expressible = Atrophic or Cicatricial MGD (exclusion at Visit 1 and 2) 0= clear secretion (normal)
  1. opaque secretion with normal viscosity
  2. opaque secretion with increased viscosity
  3. severely thickened secretion, toothpaste consistency At each time point, these characteristics will be compared to baseline at day 0.
Best corrected distance visual acuity | 2, 4 and 6 weeks
  as compared to baseline measurement at day 0
Corneal staining | 2, 4 and 6 weeks
  Using NEI industry workshop scale. Scores will be compared to baseline measurement at day 0
Axial topography based astigmatism pattern | 2, 4 and 6 weeks
  Patterns will be compared to baseline at day 0. All topography testing will be performed using the same machine and system, the Carl Zeiss Meditec Atlas, Model 9000, system 3.0.0.39.
  The topographic pattern will be reviewed by a masked investigator (masked to eye randomization), and categorized as one of the following:
  1. Normal/Symmetrical: Includes round, oval, or symmetric bowtie patterns
  2. Asymmetric bowtie: Differentiated from symmetric bowtie by a difference between axial keratometry readings along the two lobes of >1D at points 1.5mm from the center, or a difference in the widths of the lobes of the bowties at that distance of >33%.
  3. Irregular: Includes skewed radial axis (skewing by >20%), inferior or superior steepening (I-S asymmetry >1.2D); or a pattern that does not fit either 1 or 2 above.
Intraocular Lens(IOL) Master Keratometry | 2, 4 and 6 weeks
  As compared to baseline at day 0.
Change in Corneal Irregularity Measurement | 2 weeks, 6 weeks
  Topographically defined corneal smoothness as compared to baseline measurement at day 0

OTHER OUTCOMES:
Tear film break-up time | 2, 4 and 6 weeks
  Fluorescein break up time

CONTACTS AND LOCATIONS:
Overall Officials: Brad H Feldman, MD, Principal Investigator — Philadelphia Eye Associates
Locations (1):
- Philadelphia Eye Associates, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No